CLINICAL TRIAL: NCT04400318
Title: Randomized, Double Blind, Placebo Controlled Study to Evaluate the Effect of Dupilumab on Airway Inflammation Through Assessments of Lung Function, Mucus Plugging and Other Lung Imaging Parameters in Patients With Asthma
Brief Title: The Effect of Dupilumab on Lung Inflammation and Related Changes in Airway Volumes Detectable by Functional Respiratory Imaging in Patients With Moderate-severe Asthma
Acronym: VESTIGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LPS15834; U1111-1238-4679 (Registry Identifier: ICTRP); 2019-004647-74 (EudraCT Number)
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab (Experimental): Participants received a loading dose of dupilumab 600 mg as 2 subcutaneous (SC) injections on Day 1, followed by a single dupilumab 300 mg SC injection Q2W for 24 weeks along with a stable dose of medium to high ICS dose in combination with a second controller medication +/- a third controller.
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Participants received placebo matched to dupilumab as 2 x 2 mL SC injections on Day 1, followed by a single SC injection Q2W for 24 weeks along with a stable dose of medium to high ICS dose in combination with a second controller medication +/- a third controller.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — solution for injection subcutaneous
  Other Names: SAR231893 Dupixent
  Arms: Dupilumab
Drug: Placebo — Solution for injection subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

• To assess the effect of dupilumab on lung inflammation and related changes in airway volumes detectable by functional respiratory imaging

Secondary Objective:

* To evaluate the effect of dupilumab at Week 24 on bronchodynamics, hyperinflation, airway resistance, airway wall thickness, ventilation defects and mucus plugging derived from high-resolution computed tomography (HRCT) scans, patient-reported outcomes, FeNO and spirometry.
* To evaluate safety of dupilumab

DETAILED DESCRIPTION:
The study duration for each participant was a total of minimum 29 weeks and up to 41 weeks. This included 4 weeks +/-1 week screening period, 24 weeks of treatment period and a follow-up period up to 12 weeks or until the participants switched to commercialized dupilumab (or other biologic products), whatever came first.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age inclusive with the diagnosis of asthma based on Global Strategy for Asthma Management and Prevention (GINA) 2019 at the time of signing the informed consent
* History of ≥1 exacerbation(s) in the previous year
* Uncontrolled moderate to severe asthma (ACQ-5 ≥1.5) at visit (V)1 and V2, prior to randomization
* Pre-bronchodilator FEV1 ≤80% of predicted normal at V1 and V2, prior to randomization
* Exhibit bronchodilator reversibility (≥12% and 200 mL improvement in FEV1 post SABA administration) during screening, prior to randomization
* Blood eosinophil ≥300 cells /µL and FeNO ≥25 ppb during screening, prior to randomization

NOTES:

* Historical values of blood eosinophil count meeting the eligibility criterion measured within 6 months prior to SV1 in the absence of OCS treatment are allowed.
* FeNO value to be checked for eligibility at V2 as well. -Existing treatment with medium to high dose ICS in combination with a second controller (e.g. LABA, LTRA) ± a third controller. The dose regimen should be stable ≥1 month prior V1 and during screening.

Exclusion Criteria:

* Current smoker (cigarette or e-cigarette) or cessation of smoking within 1 year prior randomization
* Previous smoker with a smoking history >10 pack-years
* Known hypersensitivity to dupilumab or any of its excipients
* A subject who experiences an asthma exacerbation (defined as a deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with systemic steroids) during screening
* Current acute bronchospasm or status asthmaticus
* Diagnosed pulmonary (other than asthma) or systemic disease associated with elevated peripheral eosinophil counts
* History or clinical evidence of chronic obstructive pulmonary disease (COPD) including Asthma-COPD Overlap Syndrome (ACOS) or any other significant lung disease (eg, lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, bronchiectasis, Churg-Strauss Syndrome, etc)
* Active tuberculosis, latent untreated tuberculosis or a history of incompletely treated tuberculosis or non-tuberculous mycobacterial infection unless it is well documented by a specialist that the participants has been adequately treated and the treatment with a biologic agent can be initiated, in the medical judgment of the Investigator and/or infectious disease specialist. Tuberculosis testing would only be performed on a country by country basis according to the routine clinical practice and the local guidelines, if required by regulatory authorities or ethics committees
* History of or current evidence of clinically significant disease in any non-respiratory system (e.g. cardiovascular, hepatic, nervous system, gastrointestinal, endocrinological, rheumatological, dermatological), which, in the judgment of the Investigator, could interfere with the study or require treatment that might interfere with the study
* Current evidence of clinically significant oncological disease, which in the opinion of the investigator may interfere with the objectives of the study or put the subject at undue risk
* Participants with any of the following results at V1:

  * Positive (or indeterminate) hepatitis B surface antigen (HBs Ag) or
  * Positive Hepatitis B IgM core antibody (IgM HBc Ab) or
  * Positive total hepatitis B core antibody (total HBc Ab) confirmed by positive HBV DNA or
  * Positive hepatitis C antibody (HCV Ab) confirmed by positive HCV RNA
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at V1
* Any biologic therapy (including experimental treatments and dupilumab) or any other biologic therapy/immunosuppressant within 3 months prior to V1
* Treatment with live (attenuated) vaccine within 4 weeks before V1. For participants who have vaccination with live, attenuated vaccines planned during the course of the study (based on national vaccination schedule/local guidelines), it will be determined, after consultation with a physician, whether the administration of vaccine can be postponed until after the end of the study, or preponed to before the start of the study without compromising the health of the participant:

  * Participants for whom administration of live (attenuated) vaccine can be safely postponed would be eligible to enroll into the study.
  * Participants who have their vaccination preponed can enroll in the study only after a gap of 4 weeks following administration of the vaccine.
* Treatment with oral corticosteroids (OCS) within 2 weeks prior to V1
* Enrolled in other ongoing studies regardless of the investigational product
* Treatment with an investigational drug within 1 month or within 5 half-lives (if known), whichever is longer, prior to V1
* Suspected or high risk of parasitic infection (helminthic infection), unless clinical and (if necessary) laboratory assessments have ruled out active infection prior to randomization
* Females who are lactating, breastfeeding, or who are pregnant
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or subjects who are legally institutionalized
* Participants are dependent on the Sponsor or Investigator (in conjunction with Section 1.61 of the ICH GCP Ordinance E6)
* Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study
* Any country-related specific regulation that would prevent the subject from entering the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (10):
  - Allianz Research Institute Site Number : 8400020, Westminster, California
  - University of Kansas School of Medicine Site Number : 8400008, Kansas City, Kansas
  - University of Michigan Site Number : 8400002, Ann Arbor, Michigan
  - The Lung Research Center Site Number : 8400010, Chesterfield, Missouri
  - American Health Research Site Number : 8400005, Charlotte, North Carolina
  - Velocity Clinical Research, Medford Site Number : 8400014, Medford, Oregon
  - Medical University of South Carolina - Pulmonary & Critical Care Clinical Research Program Site Number : 8400009, Charleston, South Carolina
  - VitaLink Research-Greenville Site Number : 8400013, Greenville, South Carolina
  - VitaLink Research - Spartanburg Site Number : 8400011, Spartanburg, South Carolina
  - ~Spartanburg Medical Research Site Number : 8400004, Spartanburg, South Carolina
- Bulgaria (13):
  - Investigational Site Number : 1000013, Dupnitsa
  - Investigational Site Number : 1000004, Montana
  - Investigational Site Number : 1000018, Plovdiv
  - Investigational Site Number : 1000012, Plovdiv
  - Investigational Site Number : 1000008, Rousse
  - Investigational Site Number : 1000015, Sofia
  - Investigational Site Number : 1000005, Sofia
  - Investigational Site Number : 1000003, Sofia
  - Investigational Site Number : 1000006, Sofia
  - Investigational Site Number : 1000011, Sofia
  - Investigational Site Number : 1000010, Sofia
  - Investigational Site Number : 1000002, Sofia
  - Investigational Site Number : 1000007, Stara Zagora
- Denmark (4):
  - Investigational Site Number : 2080006, Aarhus N
  - Investigational Site Number : 2080002, Copenhagen
  - Investigational Site Number : 2080003, Copenhagen Nv
  - Investigational Site Number : 2080001, Hvidovre
- Investigational Site Number : 2500001, Montpellier, France
- Italy (3):
  - Investigational Site Number : 3800003, Cona, Ferrara
  - Investigational Site Number : 3800004, Rozzano, Milano
  - Investigational Site Number : 3800001, Pisa
- Portugal (5):
  - Investigational Site Number : 6200004, Coimbra
  - Investigational Site Number : 6200005, Guimarães
  - Investigational Site Number : 6200006, Lisbon
  - Investigational Site Number : 6200003, Porto
  - Investigational Site Number : 6200001, Porto
- Romania (6):
  - Investigational Site Number : 6420005, Bragadiru
  - Investigational Site Number : 6420008, Brasov
  - Investigational Site Number : 6420006, Cluj-Napoca
  - Investigational Site Number : 6420001, Cluj-Napoca
  - Investigational Site Number : 6420007, Oradea
  - Investigational Site Number : 6420003, Timișoara
- Saudi Arabia (6):
  - Investigational Site Number : 6820008, Dammam
  - Investigational Site Number : 6820004, Jeddah
  - Investigational Site Number : 6820006, Riyadh
  - Investigational Site Number : 6820001, Riyadh
  - Investigational Site Number : 6820002, Riyadh
  - Investigational Site Number : 6820010, Riyadh
- Spain (4):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, Santiago de Compostela, Galicia [Galicia]
  - Investigational Site Number : 7240005, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240003, Madrid, Madrid, Comunidad de
- Investigational Site Number : 7520001, Lund, Sweden
- Taiwan (4):
  - Investigational Site Number : 1580004, Kaohsiung City
  - Investigational Site Number : 1580002, Taichung
  - Investigational Site Number : 1580003, Tainan
  - Investigational Site Number : 1580001, Taipei
- Ukraine (6):
  - Investigational Site Number : 8040003, Chernivtsi
  - Investigational Site Number : 8040001, Ivano-Frankivsk
  - Investigational Site Number : 8040002, Kharkiv
  - Investigational Site Number : 8040004, Kyiv
  - Investigational Site Number : 8040005, Odesa
  - Investigational Site Number : 8040007, Ternopil
- United Kingdom (2):
  - Investigational Site Number : 8260001, Leicester, Leicestershire
  - Investigational Site Number : 8260002, Bradford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Porsbjerg C, Dunican EM, Lugogo NL, Castro M, Papi A, Backer V, Brightling CE, Bourdin A, Virchow JC, Zhang M, Soler X, Rowe PJ, Deniz Y, de Prado Gomez L, Sacks HJ, Jacob-Nara JA. Effect of Dupilumab on Mucus Burden in Patients with Moderate-to-Severe Asthma: The VESTIGE Trial. Am J Respir Crit Care Med. 2025 Oct 27. doi: 10.1164/rccm.202410-1894OC. Online ahead of print. PMID 41145399
- [Derived] Castro M, Papi A, Porsbjerg C, Lugogo NL, Brightling CE, Gonzalez-Barcala FJ, Bourdin A, Ostrovskyy M, Staevska M, Chou PC, Duca L, Pereira AM, Fogarty C, Nadama R, Zhang M, Rodrigues A, Soler X, Sacks HJ, Deniz Y, Rowe PJ, de Prado Gomez L, Jacob-Nara JA. Effect of dupilumab on exhaled nitric oxide, mucus plugs, and functional respiratory imaging in patients with type 2 asthma (VESTIGE): a randomised, double-blind, placebo-controlled, phase 4 trial. Lancet Respir Med. 2025 Mar;13(3):208-220. doi: 10.1016/S2213-2600(24)00362-X. Epub 2025 Feb 10. PMID 39947221
- See also: LPS15834 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25276&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 317 participants were screened from 20 Jun 2020 to 06 Jan 2023 at 72 study sites in 14 countries of which 208 participants were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 109 participants were randomized in a ratio of 2:1 to receive dupilumab 300 milligrams (mg) or matching placebo every 2 weeks (Q2W) for 24 weeks. Randomization was stratified by inhaled corticosteroids (ICS) dose level (medium/high no less than 40% in 'high ICS' stratum) and region (Eastern Europe/Rest of the World [ROW]).
Groups:
- Dupilumab 300 mg Q2W: Participants received a loading dose of dupilumab 600 mg as 2 subcutaneous (SC) injections on Day 1, followed by a single dupilumab 300 mg SC injection Q2W for 24 weeks along with a stable dose of medium to high ICS dose in combination with a second controller medication +/- a third controller.
- Placebo: Participants received placebo matched to dupilumab as 2 x 2 milliliter (mL) SC injections on Day 1, followed by a single SC injection Q2W for 24 weeks along with a stable dose of medium to high ICS dose in combination with a second controller medication +/- a third controller.
Period: Overall Study
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Started | 72 | 37
Completed | 70 | 33
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Not Related to Coronavirus Disease 2019 Pandemic | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) analysis set consisted of randomized participant (participant with a study intervention kit number allocated and recorded in the interactive voice recognition system [IVRS]/ interactive web response system [IWRS] database, regardless of whether the study intervention kit was used or not).
Groups:
- Dupilumab 300 mg Q2W: Participants received a loading dose of dupilumab 600 mg as 2 SC injections on Day 1, followed by a single dupilumab 300 mg SC injection Q2W for 24 weeks along with a stable dose of medium to high ICS dose in combination with a second controller medication +/- a third controller.
- Total: Total of all reporting groups
Arm/Group | Dupilumab 300 mg Q2W | Placebo | Total
Number analyzed (Participants) | 72 | 37 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (12.81) | 49.4 (12.33) | 50.4 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 22 | 68
  Male | 26 | 15 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 64 | 34 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Untrimmed Distal Specific Airway Volumes ([s]iVaw) at Total Lung Capacity (TLC) [Mean (Standard Deviation); unit: mL] — Population: Only those participants with data available at baseline are reported.
  mL
    number analyzed (Participants) | 69 | 35 | 104
    (all) | 1.90526 (0.954024) | 1.90562 (1.161739) | 1.90539 (1.022934)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Fractional Exhaled Nitric Oxide (FeNO) Less Than (<) 25 Parts Per Billion (Ppb) at Week 24
Description: FeNO was analyzed using a NIOX instrument using a flow rate of 50 milliliters per second (mL/s). This assessment was conducted prior to spirometry and following a fast of greater than or equal to (≥1) hour. The test was performed after a wash out period of bronchodilators.
Time Frame: Week 24
Population: The ITT analysis set consisted of randomized participants (participants with a study intervention kit number allocated and recorded in the IVRS/IWRS database, regardless of whether the study intervention kit was used or not).
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 72 | 37
percentage of participants | 56.9 | 10.8
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Placebo; Odds Ratio, 95% confidence interval (CI) of the odds ratio and p-value between the dupilumab and placebo group based on the Cochran-Mantel-Haenszel (CMH) test adjusted by ICS dose level (medium/high) and region (Eastern Europe/ROW); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 9.81, 95% CI 2-sided [3.13 to 30.82]

2. Primary Outcome: Percent Change From Baseline to Week 24 in Untrimmed Distal Specific Airway Volumes ([s]iVaw) at Total Lung Capacity (TLC)
Description: Specific airway volume [(s)iVaw] is the change of volume of the airways (in mL), taking into account the lung volume changes (in liter [L]) as well. It corresponds to the ratio between the airway volume (iVaw) and the lobar volume. This way the air volumes are normalized across participants and become specific. Untrimmed distal [s]iVaw at TLC was assessed based on 3-dimensional (D) rendering of high-resolution computed tomography (HRCT) scans. Baseline was defined as the last available valid (non-missing) value up to and including the day of first dose of investigational medicinal product (IMP).
Time Frame: Baseline (Day 1) to Week 24
Population: The ITT analysis set consisted of randomized participants (participants with a study intervention kit number allocated and recorded in the IVRS/IWRS database, regardless of whether the study intervention kit was used or not). Only participants with data collected at Week 24 are reported.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 68 | 34
percent change | 19.73 (8.102) | -2.04 (11.538)
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Placebo; The mixed model for repeated measures (MMRM) included study intervention, baseline value, region, ICS dose level, visits, study intervention by visit interaction, and baseline by visit interaction terms all as fixed effects. Region, ICS, study intervention and visits were considered as categorical parameters; Test type: Superiority; p = 0.138, MMRM; Least square mean difference = 21.76, 95% CI 2-sided [-7.73 to 51.25], Standard Error of Mean 14.022

3. Secondary Outcome: Change From Baseline to Week 24 in Global Lung Mucus Score (University of California, San Francisco [UCSF] Mucus Scoring)
Description: The mucus scoring system was derived, with very minor differences, from UCSF mucus score. The mucus score was calculated by counting the number of bronchopulmonary segments which contained 1 or more mucus plug, up to a maximum score of 18 corresponding to the 18 bronchopulmonary segments present in most people. In this system, a mucus plug is defined as a complete occlusion of the airway visible at TLC. Each bronchopulmonary segment is given a score of 1 (mucus plug[s] present) or 0 (mucus plug[s] absent). The segment scores of each lobe are summed to generate a total mucus score for both lungs, yielding a mucus score ranging from 0-18. Higher scores indicate worse outcome. Baseline was defined as the last available valid (non-missing) value up to and including the date of first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 68 | 34
score on a scale | -3.48 (0.463) | 1.44 (0.656)
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Placebo; MMRM model included study intervention (dupilumab, placebo), baseline value of global lung UCSF mucus scoring, region (Eastern Europe/ROW), ICS dose level (medium/high), visit (up to Week 24), study intervention-by-visit interaction and baseline-by-visit interaction as covariates; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measure is reported and continued when previous outcome measure was statistically significant at two-sided 0.05. Only 2 secondary outcome measures (#4 and #5) were included in this procedure; p < 0.001, MMRM; Least square mean difference = -4.92, 95% CI 2-sided [-6.50 to -3.34], Standard Error of Mean 0.798

4. Secondary Outcome: Percent Change From Baseline to Week 24 in Trimmed Distal Specific Airway Resistance ([s]iRaw) at TLC
Description: iRaw is defined as the total pressure drop over an airway, divided by the flow rate through that airway. The specific airway resistance (s)iRaw is derived from iRaw by multiplying the airway resistance with the lobar volume. This way, the airway resistances are normalized across participants and become specific. Trimmed distal ([s]iRaw) at TLC was assessed using HRCT scan. Baseline was defined as the last available valid (non-missing) value up to and including the day of first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 68 | 34
percent change | 36.85 (22.562) | 90.30 (32.541)
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Placebo; MMRM model included study intervention (dupilumab, placebo), baseline value of trimmed distal [s]iRaw at TLC, region (Eastern Europe/ROW), ICS dose level (medium/high), visit (up to Week 24), study intervention-by-visit interaction, and baseline-by-visit interaction as covariates; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.180, MMRM; Least square mean difference = -53.45, 95% CI 2-sided [-132.09 to 25.19], Standard Error of Mean 39.562

5. Secondary Outcome: Percent Change From Baseline to Week 24 in Untrimmed Distal Specific Airway Volumes ([s]iVaw) at Functional Residual Capacity (FRC)
Description: (s)iVaw is the change of volume of the airways (mL), taking into account the lung volume changes (in L) as well. It corresponds to the ratio between the airway volume (iVaw) and the lobar volume. Untrimmed distal [s]iVaw at FRC was assessed based on 3-D rendering of HRCT scans. Baseline was defined as the last available valid (non-missing) value up to and including the day of first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 70 | 35
percent change | 225.91 (92.250) | -17.07 (129.384)

6. Secondary Outcome: Percent Change From Baseline to Week 24 in Trimmed Distal Specific Airway Resistance ([s]iRaw) at FRC
Description: iRaw is defined as the total pressure drop over an airway, divided by the flow rate through that airway. The specific airway resistance (s)iRaw is derived from iRaw by multiplying the airway resistance with the lobar volume. This way, the airway resistances are normalized across participants and become specific. Trimmed distal [s]iRaw at FRC was assessed using HRCT scan. Baseline was defined as the last available valid (non-missing) value up to and including the day of the first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 69 | 35
percent change | 98.73 (70.143) | 207.87 (98.445)

7. Secondary Outcome: Percent Change From Baseline to Week 24 in Global Lung Lobar Volumes (iVlobes) at TLC
Description: The lung volume was determined from the HRCT scan at TLC, by identifying and grouping the voxels that represent the air in the lungs. The total lung volume along with the volume of each lobe individually was determined which allowed to pick up substantial regional physiological changes of the airways and the lobe volumes. Baseline was defined as the last available valid (non-missing) value up to and including the day of first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 68 | 34
percent change | -0.98 (1.691) | -3.74 (2.401)

8. Secondary Outcome: Change From Baseline to Week 24 in HRCT-Based Internal Airflow Distribution (IAD) for Each Lung Zone
Description: The IAD was assessed in the upper and lower lung using HRCT scan. By segmenting the lobes at FRC and TLC for each participant, the participant-specific airflow distribution can be established by assessing lobar and volume expansion. Baseline was defined as the last available valid (non-missing) value up to and including the date of the first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of IAD
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 67 | 34
percentage of IAD
  Upper Lung | -0.61 (0.803) | -0.11 (1.133)
  Lower Lung | 0.61 (0.803) | 0.11 (1.133)

9. Secondary Outcome: Change From Baseline to Week 24 in Image-Based Ventilation/Perfusion (iV/Q) at TLC for Each Lung Zone
Description: Blood vessel density can be considered a surrogate for perfusion, hence image-based perfusion (IQ) is calculated by blood vessel density at TLC multiplied by image-based volume at TLC. Image-based ventilation (IV) is calculated by the imaged volume at TLC subtracted from the image-based volume at FRC. The ventilation/perfusion ratio IV/Q is then the ratio IV/IQ. The iV/Q was assessed in the upper and lower lung using HRCT scan at TLC. Baseline was defined as the last available valid (non-missing) value up to and including the day of the first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 67 | 34
Ratio
  Upper Lung | 1.42 (0.538) | -0.45 (0.758)
  Lower Lung | 1.75 (0.579) | -0.91 (0.817)

10. Secondary Outcome: Change From Baseline to Week 24 in FeNO
Description: FeNO was analyzed using a NIOX instrument using a flow rate of 50 mL/s. This assessment was conducted prior to spirometry and following a fast of ≥1 hour. The test was performed after a wash out period of bronchodilators. Baseline was defined as the last available valid (non-missing) value up to and including the day of the first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: parts per billion
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 72 | 37
parts per billion | -35.49 (2.440) | -12.56 (3.444)

11. Secondary Outcome: Change From Baseline to Week 24 in Pre-Bronchodilator and Post-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration. Lung function parameters: pre- and post-bronchodilator FEV1 were measured by spirometry before IMP administration. Spirometry was performed after a wash out period of bronchodilators. Post-BD FEV1 was measured within 30 minutes after short-acting beta-2 agonists (2 to up to 4 puffs of albuterol/salbutamol) administration. Baseline was defined as the last available valid (non-missing) value up to and including the date of the first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 72 | 37
liter
  Pre-Bronchodilator FEV1 | 0.655 (0.0637) | 0.274 (0.0885)
  Post-Bronchodilator FEV1 | 0.468 (0.0661) | 0.151 (0.0928)

12. Secondary Outcome: Change From Baseline to Week 24 in 7 Item Asthma Control Questionnaire (ACQ-7)
Description: The ACQ-7 comprises of 7 items:first 5 items assess most common asthma symptoms: 1. frequency in past week awoken by asthma during the night; 2. severity of asthma symptoms in the morning; 3. limitation of daily activities due to asthma; 4. shortness of breath due to asthma; and 5. wheeze; plus questions 6. short-acting bronchodilator use; and 7. FEV1 (pre-bronchodilator use, % and % predicted use).Participants are asked to recall how their asthma has been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6=maximum impairment).Clinic staff scores the FEV1% predicted on a 7-point scale.A global score is calculated: the questions are equally weighted, and the overall ACQ-7 score is the mean of the 7 questions and, therefore, between 0 (totally controlled) and 6 (severely uncontrolled).Higher score indicates lower asthma control. Baseline=last available valid (non-missing) value up to and including day of the first dose of IMP.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 70 | 36
score on a scale | -1.36 (0.101) | -0.62 (0.143)

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and Adverse Events of Special Interest (AESIs)
Description: AE: any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs: AEs that developed or worsened or became serious during the TEAE period, defined as the time from the first administration of the IMP (on Day 1) to the last administration of the IMP + 98 days and up to the end of the study follow-up. Serious adverse events (SAE): AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. AESI: AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor is required.
Time Frame: From first dose of study drug (Day 1) up to end of study (up to 36 weeks)
Population: The safety analysis set included all randomized participants who received at least 1 injection of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab 300 mg Q2W | Placebo
Number analyzed (Participants) | 72 | 37
Participants
  Any TEAE | 31 | 21
  Any TESAE | 3 | 1
  Any AESI | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to end of study (up to 36 weeks)
Description: Analysis was performed on safety analysis set.
Arm/Group | Dupilumab 300 mg Q2W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/37
Serious Adverse Events (participants affected / at risk) | 3/72 | 1/37
Other Adverse Events (participants affected / at risk) | 18/72 | 15/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg Q2W (N=72) | Placebo (N=37)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eosinophilic Granulomatosis With Polyangiitis (Immune system disorders) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg Q2W (N=72) | Placebo (N=37)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Injection Site Reaction (General disorders) | 4 (10) | 1 (2)
Covid-19 (Infections and infestations) | 7 (7) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (6) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT04400318/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT04400318/SAP_001.pdf